CLINICAL TRIAL: NCT00978107
Title: A Phase I, Open-label, Dose-escalating Study of the Safety or Percutaneous Intra-tumoral Injection of TG4023 (MVA-FCU1) Combined With Systemic Administration of 5-fluorocytosine in Patients With Primary or Secondary Hepatic Tumors.
Brief Title: Trial of TG4023 Combined With Flucytosine in Liver Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG4023.01; Eudra CT 2008-005024-90
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic tumors; Metastatic colorectal cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms | interventions — Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MVA-FCU1, flucytosine — 1. TG4023: single IT injection; possibility to re-administer once,
     * Percutaneous IT injections, under radiological or ultrasound imaging guidance
     * Dose-escalating schedule of administration: 107 pfu (Cohort #1), 108 pfu (Cohort #2) and 4x108 pfu (Cohort #3),
     * MTD injected to up to 3 different lesions (Cohort #4)
  2. 5-FC (5-fluorocytosine)/flucytosine
     * Dose and dosing schedule:
       * Daily starting dose of 200 mg/kg; daily dose will be adjusted after measurement of 5-FC plasma concentration at steady state, which should be kept below 100 mg/L
       * Duration: 2 weeks.
     * Possible routes of administration:
       * PO: 500 mg tablets, qid
       * IV: 1% 250 mL vials, 45-minute infusions.
  Other Names: 5-FC

SUMMARY:
This trial is a phase I, open-label, dose-escalating study of the safety or percutaneous intra-tumoral injection of TG4023 (MVA-FCU1) combined with systemic administration of 5-fluorocytosine in patients with primary or secondary hepatic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced disease without any other standard of care treatment options:

  * hepatic metastases of colorectal cancer (CRC) or of other cancers
  * Hepatocellular carcinoma (HCC)
* At least one unresectable target tumor located in the liver, measuring 2-5 cm and accessible to IT administration of TG4023 and amenable to radiological measurement using RECIST,
* Weight ≤ 100 kg,
* Patients with stable disease, who have to discontinue chemotherapy because of intolerance,
* ECOG performance status ≤ 2,
* Life expectancy ≥ 3 months,
* Hematology:

  * Absolute neutrophil count > 1,500/mm3,
  * Hemoglobin > 9g/dL,
  * Platelet count > 100,000/mm3,
  * Prothrombin time international normalized ratio (INR) ≤ 2; partial thromboplastin time ≤ 1.66 times upper limit of normal (ULN),
* Biochemistry:

  * Total bilirubin ≤ 3 x ULN,
  * Aspartate amino-transferase (AST), alanine amino-transferase (ALT), alkaline phosphatase

    * 5.0 x ULN,
  * Creatinin clearance ≥ 40 mL/min,
  * Total albumin ≥ 30 g/L,
* Anti-vitamin K anticoagulants should have been switched for low-molecular weight heparin prior to TG4023 injection,
* Signed, written Independent Ethics Committee (IEC)-approved informed consent.

Exclusion Criteria:

* Child-Pugh stage C hepatic insufficiency,
* Impaired renal function (creatinin clearance < 40 mL/min),
* Known deficiency in dihydropyrimidine dehydrogenase (DPD) or total DPD deficiency diagnosed at baseline in those patients not previously treated with 5-FU-related compounds,
* Ascites,
* Brain metastases,
* Significant impairment of gastro-intestinal (GI) tract absorption capacity, such as total gastrectomy, gastric mucosal atrophy, extensive intestinal resections or malabsorption disease will not be treated by oral 5-FC,
* History of bleeding disorders,
* Pregnant or breast-feeding women,
* Human Immunodeficiency Virus (HIV) positive,
* Chronic use of immunodepressants within 4 weeks prior to TG4023 injection or immune-depressed patients,
* Hypersensitivity to 5-FC,
* Hypersensitivity to egg proteins,
* Concomitant or previous chemotherapy or targeted therapy within 4 weeks prior to TG4023 injection and last treatment with bevacizumab (Avastin®) within 2 months prior to TG4023 injection,
* Concomitant treatment with anti-inflammatory drugs: systemic cortico-steroids and non-steroidal anti-inflammatory drugs (NSAIDs),
* Prior gene therapy,
* Prior participation in any other research protocol involving an IMP within 2 months prior to TG4023 injection,
* Major surgery within 6 weeks of TG4023 injection,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose | 6 months

SECONDARY OUTCOMES:
Tumor response of injected and non-injected lesions Viral dissemination Proof of concept: 5-FU concentration in plasma and in tumors | 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpitaux Civils de Colmar, Colmar
  - Institut Paoli Calmette,, Marseille
  - Hôpitaux Civils de Lyon,, Pierre-Bénite
  - Centre René Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Background] Erbs P, Findeli A, Kintz J, Cordier P, Hoffmann C, Geist M, Balloul JM. Modified vaccinia virus Ankara as a vector for suicide gene therapy. Cancer Gene Ther. 2008 Jan;15(1):18-28. doi: 10.1038/sj.cgt.7701098. Epub 2007 Nov 9. PMID 17992203
- [Derived] Husseini F, Delord JP, Fournel-Federico C, Guitton J, Erbs P, Homerin M, Halluard C, Jemming C, Orange C, Limacher JM, Kurtz JE. Vectorized gene therapy of liver tumors: proof-of-concept of TG4023 (MVA-FCU1) in combination with flucytosine. Ann Oncol. 2017 Jan 1;28(1):169-174. doi: 10.1093/annonc/mdw440. PMID 28177438